CLINICAL TRIAL: NCT02405598
Title: Evaluation of Salbutamol as an Adjuvant Therapy for Pompe Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Hsiao Sang Chu, MD, MD, PhD, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201308031MINC
Record Dates: First submitted 2015-03-22; First posted 2015-04-01 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Salbutamol (Experimental): 1. age 2-6 year: 0.1mg/kg tid x 2 weeks, then gradually increase to 0.2mg/kg tid (daily total maximal12mg)
  2. age 6-12 year: 2mg tid x 2 weeks, then gradually increase to 4mg tid (daily total maximal 24mg)
  3. age 12 year and above: 4mg tidx 2 weeks, then gradually increase to 8mg tid (daily total maximal 32mg)
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Salbutamol — 1. Albuterol Syrup (1mL= Salbutamol 0.4mg, 60ml/bot)
  2. VENTOLIN TABLETS 2MG (SALBUTAMOL SULPHATE)

SUMMARY:
evaluate if beta 2-adrenergic agonist can have adjuvant effect to patients with infantile-onset Pompe disease under enzyme replacement therapy

ELIGIBILITY:
Inclusion Criteria:

1. Confirm diagnosis as Pompe disease
2. age 2 years or above
3. under at least 1 year regular recombinant human acid alpha glucosidase, and no dosage/frequency change in recent 3 months
4. Provide inform consent

Exclusion Criteria:

1. chronic heart disease such as arrhythmia, cardiomyopathy, cardiac infarction
2. history of seizure
3. history of diabetes mellitus
4. history of hyperthyroidism
5. hypokalemia
6. pregnant
7. allergy to β-agonists
8. under medications including diuretics, digoxin, beta-blockers, etc

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
10% decrement of creatinine kinase | 6 months
  measure and compare serum creatinine kinase levels
Improvement in 6-minutes walk test | 6 months
  measure and compare 6-minutes walk test

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan